CLINICAL TRIAL: NCT01486420
Title: Open Surgery Versus Ultrasound Guided Local Corticosteroid Injections in Treatment of Trigger Finger - a Randomized Controlled Trial.
Brief Title: Open Surgery Versus Corticosteroid Injections in Treatment of Trigger Finger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeppe Lange, MD (Other)
Responsible Party: Sponsor-Investigator, Jeppe Lange, MD, Senior project superviser, Regionshospitalet Silkeborg
Organization: Regionshospitalet Silkeborg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20110157
Record Dates: First submitted 2011-12-01; First posted 2011-12-06 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Trigger Finger
Keywords: Quinell grade; Open surgery; corticosteroid injections; randomized controlled trial; Trigger finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open surgery (Active Comparator)
  Interventions: Procedure: Open surgery
- Corticosteroid Injection (Active Comparator)
  Interventions: Procedure: Corticosteroid injections

INTERVENTIONS:
Procedure: Corticosteroid injections — Corticosteroid injections in and around A1-pulley.
  Arms: Corticosteroid Injection
Procedure: Open surgery — Open A1-pulley release
  Arms: Open surgery

SUMMARY:
The purpose of the study is to investigate which strategy is superior in trigger finger Quinell grade IIb-V; conventional open surgery or ultrasound guided corticosteroid injections.

ELIGIBILITY:
Inclusion Criteria:

* Trigger finger Quinell grade IIb-V in digit I-V

Exclusion Criteria:

* Former treatment of Trigger finger in affected digit
* Dupuytrens contracture in affected digit
* Allergies or intolerance to used medications
* Rheumatoid Arthritis
* Insulin dependent Diabetes Mellitus
* Amyloidosis
* Mucopolysaccharidosis
* Already included in study with another digit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quinell grade | 12 months
  Dicotomized outcome defined as +/- failure. Failure defined as Quinell grade equal to or above IIb.
  Quinell grade defined as: I Normal movement, IIa normal movement with pain/tenderness to A1-pulley, IIb anamnestic triggering but not evident at clinical exam, III triggering without locking, IV triggering with locking but actively correctable, V Locked digit, passive correctable only.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) score | 12 weeks
  Pain following either procedure measured by NRS (score 0-10, 10 is severe pain)
infection | 12 weeks
  Infection occurence following either procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe Lange, M.D., Study Director — Center for Planned Surgery - Regionalhospital Silkeborg
Locations (1):
- Center for Planned surgery - Regionalhospital Silkeborg, Silkeborg, Denmark

REFERENCES:
- [Derived] Hansen RL, Lange J. Surgery versus ultrasound-guided steroid injections for trigger finger disease: protocol of a randomized controlled trial. Dan Med J. 2013 May;60(5):A4633. PMID 23673265